CLINICAL TRIAL: NCT03957642
Title: Diagnostic Value of Systematic Imaging Examination in Embedded Optic Disc Drusen in Adolescents With Mild Visual Impairment
Brief Title: Systematic Imaging Examination in ODD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiang Zhu, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: Systematic Imaging Examination
Record Dates: First submitted 2019-05-19; First posted 2019-05-21 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Optic Disk Drusen
MeSH Terms: conditions — Optic Disk Drusen

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the diagnostic value of systematic ophthalmologic imaging examination in the diagnosis of embedded optic disc drusen (ODD) in adolescents with mild visual impairment.

DETAILED DESCRIPTION:
Patients are evaluated through optometric examination, fundus photography, visual field examination, OCT, US, and FFA.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Age 14-28.
3. The results of visual acuity examination suggest mild visual impairment.
4. The results of ophthalmologic examination showed that the blurred degree of the local boundary of the optic disc was different and the optic disc was congested.

Exclusion Criteria:

1. patients with amblyopia.
2. patients with neurological disease.

Ages: 14 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents with mild visual impairment accompanied by disc flushing, crowded optic disc, and a blurred disc halo.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
detection rate of embedded ODD | 1 week
  detection rate of embedded ODD

CONTACTS AND LOCATIONS:
Overall Officials: Xiuhua Jia, Dorctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The third affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China